CLINICAL TRIAL: NCT03559569
Title: Impact of Endothelial and Leukocyte Senescence in Circulatory Shock States
Acronym: Seneshock
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7031
Record Dates: First submitted 2018-05-17; First posted 2018-06-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Shock; Cardiovascular Diseases; Infection
Keywords: Shock; Cardiovascular Diseases; Infection
MeSH Terms: conditions — Shock; Cardiovascular Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Only whole blood will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with circulatory shock: 500 patients with circulatory shock hospitalize in ICU will be prospectively included to assess the effect of this pathology on the senescence phenotype
  Interventions: Biological: Biological samples will be done to evaluate the endothelial and leukocyte senescence.
- Healthy volunteers: 20 healthy volunteers will be included to assess the effect of no pathology on the senescence phenotype.
  Interventions: Biological: Biological samples will be done to evaluate the endothelial and leukocyte senescence.

INTERVENTIONS:
Biological: Biological samples will be done to evaluate the endothelial and leukocyte senescence. — Noninvasive, reproducible, and sensitive methods to measure cardiac function, endothelial function, and arterial stiffness will be assess.

SUMMARY:
Circulatory shocks (CS) are life-threatening, acute organ dysfunction. Advances in critical care medicine have decreased early hospital mortality, increasing the number of surviving patients. Regrettably, these survivors are at increased risk of new infections but also of cardiovascular disease.

The investigators hypothesize that CS with multi-organ dysfunction is associated with premature senescence of endothelial cells and immune cells and promotes endothelial thrombogenicity and immunosenescence leading to cardiovascular disease and secondary infections.

The aim of this work is therefore to evaluate the contribution of endothelial and leucocytes senescence to the occurrence of secondary events (infectious and cardiovascular) in patients with a CS. It will provide a better understanding of the pathogenesis of cardiovascular and immune diseases following a CS, likely to guide new management strategies to prevent their occurrence.

ELIGIBILITY:
Inclusion criteria:

* Circulatory shock
* patient with health care insurance

Exclusion criteria:

* Patients' refusal to participate in clinical research
* Pregnant woman
* Breastfeeding woman
* A patient with a protective order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the intensive care unit of the "Nouvel Hôpital Civil de Strasbourg" for a circulatory shock will be included.
  Healthy volunteer will be included in our Clinical Investigation Center of the "Hôpitaux Universitaires de Strasbourg"
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The main criterion will be the acquisition of a senescent phenotype concerning leukocytes and endothelial cells. | 1 year
  Biological samples will be done to evaluate the endothelial and leukocyte senescence.

SECONDARY OUTCOMES:
Incidence of cardiovascular events and secondary infection in hospitalized patients in intensive care unit for circulatory shock states | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ferhat MEZIANI, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Service de Réanimation médicale du NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chomel L, Vogt M, Demiselle J, Le Borgne P, Tschirhart M, Morandeau V, Merdji H, Miguet L, Helms J, Meziani F, Mauvieux L. TLRs1-10 Protein Expression in Circulating Human White Blood Cells during Bacterial and COVID-19 Infections. J Innate Immun. 2024;16(1):216-225. doi: 10.1159/000536593. Epub 2024 Mar 8. PMID 38461810